CLINICAL TRIAL: NCT05446454
Title: Criterion and Convergent Validity of Activity Monitors to Study Walking Activity
Brief Title: Validity of Activity Monitors to Study Walking
Acronym: VAMOS
Status: Completed | Type: Observational
Sponsor: University of Rennes 2 (Other)
Collaborators: Ecole normale supérieure de Rennes (FRANCE) (Unknown)
Responsible Party: Principal Investigator, Alexis LE FAUCHEUR, Associate professor, University of Rennes 2
Other Study IDs: 2020-A03382-37
Record Dates: First submitted 2022-03-30; First posted 2022-07-06 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Validity Study of Activity Monitors in Healthy Subjects
Keywords: criterion validity; convergent validity; wearable activity monitors; (intermittent) walking; physical activity bouts; energy expenditure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Wearable activity monitors represent a real opportunity to assess people' daily walking activity, however their level of validity remains poorly understood in the assessment of intermittent walking activity, i.e. as it occurs in everyday life conditions. Indeed, the available validation studies mainly focused on steps count accuracy of wearable activity monitors, but their validity to detect and quantify bouts of intermittent walking in daily life conditions remains insufficiently studied. It is important not only to determine which indicators would be the most accurate but also which methods would be the most suitable for detecting intermittent walking bouts, and then estimating energy expenditure. The main objective of the VAMOS project is to study the criterion and convergent validity of consumer-level and research-grade wearable activity monitors in assessing daily life intermittent walking in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 20 years old and under 80 years old.
* Have understood the objectives of the study and its constraints.
* Have read and signed a free and informed consent.
* Be affiliated to the French social security system

Exclusion Criteria:

* Known contraindications or limitations to walking, and reported by the participant.
* Case of hypertension, heart failure, angina pectoris, diabetes, chronic obstructive pulmonary disease, proven by the presence of medication in relation to these diseases and the medical history reported by the participant.
* Case of factors, medical treatments, or diseases likely to lead to a functional limitation to walking and/or a significant modification of the physiological responses to exercise, e.g. active smoking (ongoing or weaned for less than six months), cancer (ongoing), Parkinson's disease, kidney failure (ongoing), proven by the presence of medication in relation to these diseases and the medical history reported by the participant.
* History of cardiovascular disease (heart failure, stroke, heart attack myocardium…) reported by the participant.
* Woman with known ongoing pregnancy (self-declared) or breastfeeding woman.
* Adults subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.
* Simultaneous participation in another research involving the human person.
* Consent withdrawal during the study.
* Any health concern that would appear during the study and that no longer would allow the person to continue to participate.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy participants aged between 20-80 years old will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Detection rate of daily life walking bouts | 8 days
  Detection rate of daily life walking bouts by wearable activity monitors
Error level in the estimation of walking energy expenditure | 1 day
  Error level in the estimation of walking energy expenditure by wearable activity monitors

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Le Faucheur, Principal Investigator — Ecole normale supérieure de Rennes (FRANCE)
Locations (1):
- Health, Sport and Movement Laboratory (M2S), Bruz, France